CLINICAL TRIAL: NCT00784095
Title: Outlook: An Intervention to Improve Quality of Life in Serious Illness
Brief Title: Outlook Quality of Life Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: IAD 07-162
Record Dates: First submitted 2008-10-30; First posted 2008-11-03 (Estimated); Results first posted 2016-03-22 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Cancer; Congestive Heart Failure; Chronic Obstructive Pulmonary Disease
Keywords: quality of life
MeSH Terms: conditions — Neoplasms; Heart Failure; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Preparation and Completion (Experimental): Subjects in the first group ("treatment") met with the facilitator three times for a period of forty-five minutes to one hour to discuss issues of life completion and preparation. In the first session, subjects were asked to discuss issues related to life review. In session two, participants spoke about issues of regret and forgiveness. In the final session, subjects discussed issues of heritage and legacy.
  Interventions: Other: Life completion and preparation
- Attention Control (Active Comparator): The subjects in the second group ("attention control") met with a facilitator three times for 45 minutes and listened to a non-guided relaxation CD.
  Interventions: Other: Attention Control
- True Control (No Intervention): Subjects in the third group ("true control") were exposed to no intervention or attention control.

INTERVENTIONS:
Other: Life completion and preparation — Subjects will discuss life review, issues of forgiveness and heritage and legacy.
  Arms: Preparation and Completion
Other: Attention Control — Subjects will listen to a non-guided relaxation CD.
  Arms: Attention Control

SUMMARY:
The purpose of this study is to determine whether discussions of life story, forgiveness, and future goals improve quality of life for patients with serious illness.

DETAILED DESCRIPTION:
This is a pilot randomized control trial to evaluate the feasibility of the Outlook intervention. 36 veterans with advanced cancer, congestive heart failure (CHF) or chronic obstructive pulmonary disease (COPD) will be randomly assigned to one of three intervention groups and complete a brief battery of pre-test measures. Subjects in the first group ("treatment") will meet with a facilitator three times for a period of 45 min-1 hour. In the first session, subjects will be asked to discuss issues related to life review. In the second session, participants will be asked to speak in more depth about issues such as regret, forgiveness and things left undone, In the final session, subjects will focus on heritage and legacy. The subjects in the second group ("attention control") will meet with a facilitator three times for a period of 45 min- 1 hour and listen to a non-guided relaxation compact disk (CD). The third group of participants ("true control") will be exposed to no intervention or attention control. One week and two weeks later, participants in all groups will receive post-test measures administered by a blinded interviewer.

ELIGIBILITY:
Inclusion Criteria:

Patients with advanced cancer, CHF or COPD.

Exclusion Criteria:

Cognitive impairment, inability to speak, non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-12; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen E. Steinhauser, PhD, Principal Investigator — Durham VA Medical Center HSR&D COE
Locations (1):
- Durham VA Medical Center HSR&D COE, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sautter JM, Tulsky JA, Johnson KS, Olsen MK, Burton-Chase AM, Lindquist JH, Zimmerman S, Steinhauser KE. Caregiver experience during advanced chronic illness and last year of life. J Am Geriatr Soc. 2014 Jun;62(6):1082-90. doi: 10.1111/jgs.12841. Epub 2014 May 6. PMID 24803020

RESULTS

PARTICIPANT FLOW:
Groups:
- Preparation and Completion: Subjects in the first group ("treatment")will meet with the facilitator three times for a period of forty-five minutes to one our. In the first session, subjects will be asked to discuss issues related to life review. In session two, participants will speak about issues of regret and forgiveness. In the final session, subjects will focus on heritage and legacy.
  Life completion and preparation: Subjects will discuss life review, issues of forgiveness and heritage and legacy.
- Attention Control: The subjects in the second group ("attention control") will meet with a facilitator three times for 45 minutes and listen to a non-guided relaxation CD.
  Attention Control: Subjects will listen to a non-guided relaxation CD.
- True Control: Subjects in the third group ("true control") will be exposed to no intervention or attention control.
Period: Overall Study
Arm/Group | Preparation and Completion | Attention Control | True Control
Started | 12 | 12 | 12
Completed | 12 | 11 | 11
Not Completed | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Preparation and Completion | Attention Control | True Control | Total
Number analyzed (Participants) | 12 | 12 | 12 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (10) | 68 (10) | 69 (14) | 67 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 0 | 1
  Male | 12 | 11 | 12 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 5 | 4 | 14
  White | 7 | 5 | 5 | 17
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 12 | 36

OUTCOME MEASURES:

1. Primary Outcome: Quality of Life - Preparation
Description: Quality Of Life At The End Of Life (the QUAL-E 2009) is a 31 item measure of quality of life at the end of life assessing five domains: life completion, relationship with health care providers, preparation for death, physical symptoms and affective social support. The 4-item preparation sub-scale is a primary outcomes measure with each item scaled from 1 to 5 with a minimum of 5, maximum of 20 score with higher scores indicating better preparation.
Time Frame: Baseline, 6 and 8 week follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Preparation and Completion | Attention Control | True Control
Number analyzed (Participants) | 12 | 11 | 11
units on a scale
  Baseline | 14.4 (3.9) | 16.0 (3.7) | 15.4 (4.4)
  6 week follow up | 15.2 (3.8) | 14.8 (5.1) | 14.5 (3.9)
  8 week follow up | 16.3 (2.7) | 16.1 (4.6) | 14.5 (4.4)
Statistical Analysis 1: Comparison: Preparation and Completion vs True Control; Intervention (Preparation and Completion) versus True Control at 8 weeks; Test type: Superiority or Other; p = .047, Mixed Models Analysis; Mean Difference (Final Values) = 2.9, 95% CI 2-sided [.04 to 5.7]
Statistical Analysis 2: Comparison: Preparation and Completion vs Attention Control; Intervention (Preparation and Completion) versus Attention Control at 8 weeks; Test type: Superiority or Other; Mean Difference (Final Values) = 1.8, 95% CI 2-sided [-1.1 to 4.7]

2. Secondary Outcome: Functional Status ADL
Description: Rosow-Breslau Activities of Daily Living scale range 17-51 with higher scores indicating greater ability.
Time Frame: Baseline, 6 and 8 week follow ups
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Preparation and Completion: Subjects in the first group ("treatment")met with the facilitator three times for a period of forty-five minutes to one hour to discuss issues of life completion and preparation. In the first session, subjects were asked to discuss issues related to life review. In session two, participants spoke about issues of regret and forgiveness. In the final session, subjects discussed issues of heritage and legacy.
  Life completion and preparation: Subjects will discuss life review, issues of forgiveness and heritage and legacy.
Arm/Group | Preparation and Completion | Attention Control | True Control
Number analyzed (Participants) | 12 | 11 | 11
units on a scale
  Baseline | 22.3 (4.4) | 21.0 (2.3) | 29.7 (6.4)
  6 week follow up | 23 (5.7) | 24 (8.1) | 30.6 (8.2)
  8 week follow up | 23.1 (5.3) | 21.8 (4.0) | 29.8 (8.0)
Statistical Analysis 1: Comparison: Preparation and Completion vs True Control; Intervention (Preparation and Completion) versus True Control at 8 weeks; Test type: Superiority or Other; Mean Difference (Final Values) = 1.2, 95% CI 2-sided [-3.2 to 5.6]
Statistical Analysis 2: Comparison: Preparation and Completion vs Attention Control; Intervention (Preparation and Completion) versus Attention Control at 8 weeks; Test type: Superiority or Other; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-5.6 to 3.3]

3. Secondary Outcome: Center for Epidemiology Studies - Depression Scale (CES-D)
Description: Center for Epidemiology Studies - Depression Scale (CES-D) is a 10-item measure of depression. Items are rated on a 4 point likert scale with total scores ranging from 0-30. Higher scores indicate greater depressive symptoms.
Time Frame: Baseline, 6 and 8 week follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Preparation and Completion | Attention Control | True Control
Number analyzed (Participants) | 12 | 11 | 11
units on a scale
  Baseline | 12.0 (5.0) | 12.0 (8.3) | 13.4 (6.6)
  6 week follow up | 12.4 (5.4) | 12.6 (7.7) | 12.3 (6.8)
  8 week follow up | 9.4 (4.2) | 12.5 (8.9) | 12.1 (5.9)
Statistical Analysis 1: Comparison: Preparation and Completion vs True Control; Intervention (Preparation and Completion) versus True Control at 8 weeks; Test type: Superiority or Other; Mean Difference (Final Values) = -1.6, 95% CI 2-sided [-6.2 to 2.9]
Statistical Analysis 2: Comparison: Preparation and Completion vs Attention Control; Intervention (Preparation and Completion) versus Attention Control at 8 weeks; Test type: Superiority or Other; Mean Difference (Final Values) = -3.6, 95% CI 2-sided [-8.2 to 1.0]

4. Secondary Outcome: POMS Anxiety Sub-scale
Description: The anxiety sub-scale from the modified Brief Profile of Mood States (POMS) is a 5-item measure of psychological distress.Items are on a 5-point likert scale with scoring ranging from 5-25. Higher scores indicate greater anxiety.
Time Frame: Baseline, 6 and 8 week follow ups
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Preparation and Completion | Attention Control | True Control
Number analyzed (Participants) | 12 | 11 | 11
units on a scale
  Baseline | 5.0 (5.5) | 4.1 (4.1) | 5.3 (4.4)
  6 week follow up | 5.1 (4.9) | 5.0 (4.0) | 5.9 (4.4)
  8 week follow up | 4.6 (3.3) | 4.8 (5.4) | 5.3 (4.2)
Statistical Analysis 1: Comparison: Preparation and Completion vs True Control; Intervention (Preparation and Completion) versus True Control at 8 weeks; Test type: Superiority or Other; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-4.5 to 3.4]
Statistical Analysis 2: Comparison: Preparation and Completion vs Attention Control; Intervention versus Attention Control at 8 weeks; Test type: Superiority or Other; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-5.1 to 3.0]

5. Primary Outcome: QUAL-E Completion Sub-scale
Description: A sub-scale of the QUAL-E quality of life at the end of life measures. The scale range was 5-35 with higher scores indicating more positive sense of completion.
Time Frame: Baseline, 6 and 8 week follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Preparation and Completion | Attention Control | True Control
Number analyzed (Participants) | 12 | 11 | 11
units on a scale
  Baseline | 22.4 (6.5) | 24.5 (5.2) | 22.5 (6.9)
  6 week follow up | 22.6 (5.6) | 25.3 (5.2) | 23.1 (6.1)
  8 week follow up | 23.4 (5.6) | 24.1 (5.9) | 24.4 (7.7)
Statistical Analysis 1: Comparison: Preparation and Completion vs True Control; Intervention (Preparation and Completion) versus True Control at 8 weeks; Test type: Superiority or Other; Mean Difference (Final Values) = -.6, 95% CI 2-sided [-4.8 to 3.7]
Statistical Analysis 2: Comparison: Preparation and Completion vs Attention Control; Intervention (Preparation and Completion) versus Attention Control at 8 weeks; Test type: Superiority or Other; Mean Difference (Final Values) = 2.4, 95% CI 2-sided [-1.9 to 6.7]

ADVERSE EVENTS:
Groups:
- Preparation and Completion: Subjects in the first group ("treatment") met with the facilitator three times for a period of forty-five minutes to one our. In the first session, subjects were asked to discuss issues related to life review. In session two, participants spoke about issues of regret and forgiveness. In the final session, subjects focused on heritage and legacy.
  Life completion and preparation: Subjects will discuss life review, issues of forgiveness and heritage and legacy.
- Attention Control: The subjects in the second group ("attention control") met with a facilitator three times for 45 minutes and listen to a non-guided relaxation CD.
  Attention Control: Subjects listened to a non-guided relaxation CD.
Arm/Group | Preparation and Completion | Attention Control | True Control
Serious Adverse Events (participants affected / at risk) | 0/12 | 1/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Preparation and Completion (N=12) | Attention Control (N=12) | True Control (N=12)
Death (General disorders) | 0 (0) | 1 (1) | 0 (0) — All patients in the trial were had advanced life-limiting illness. This was deemed not to be an unexpected event.

LIMITATIONS AND CAVEATS:
Therefore, due to the small sample size, finding are met with caution. Subjects were not randomized by any condition. As a result, those in the Control arm were more functionally able than the other two arms at baseline.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No